## STUDY PROTOCOL

Use of transcutaneous electrical nerve stimulation (TENS) for the recovery of oral function after orthognathic surgery

NCT ID not yet assigned

05/11/2020

## Statistical analysis

Descriptive statistics will be conducted to calculate distributions, frequencies, means and standard deviations for sex, malocclusion, and the results for maximum opening, bite force, inflammation, and pain in each group (experimental and control).

The Kolmogorov-Smirnov test will be applied to check the normality of variable distributions and Levene's test to check the equality of variances.

The Student's t-test will be employed to evaluate the difference in each measurement between experimental and control groups.

The paired Student's t-test will be used to compare measurements before and after TENS/sham-TENS in the same patient.

The GLM repeated-measures procedure will be applied to analyze the results for each group over time.

SPSS 22.0 ® for Windows will be used for statistical analysis

P≤0.05 was considered significant in all tests.